CLINICAL TRIAL: NCT07368634
Title: An Exploratory Clinical Study of EBV-TCR-T Cell Injection for the Treatment of EBV DNAemia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Exploratory Study of EBV-TCR-T Cell Injection for EBV DNAemia After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daihong Liu (Other)
Responsible Party: Sponsor-Investigator, Daihong Liu, Director, Department of Hematology, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2025-797
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Epstein-Barr Virus Infection; Post-Transplant Lymphoproliferative Disorder
Keywords: EBV DNAemia; TCR-T Cell Therapy; Dose Escalation Study
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV-TCR-T Cell Injection (Experimental): Participants enrolled in this arm will receive EBV-specific T cell receptor-engineered T cells (EBV-TCR-T cell injection) administered by intravenous infusion. EBV-TCR-T cells are genetically modified T lymphocytes designed to recognize and eliminate Epstein-Barr virus-infected cells.
  Participants will receive EBV-TCR-T cell infusions at predefined dose levels according to the study protocol. Infusions are administered weekly, with up to three infusions given on Day 0, Day 7, and Day 14, depending on safety and virologic response. Safety, tolerability, and preliminary efficacy will be evaluated throughout the study.
  Interventions: Biological: EBV-TCR-T Cell Injection

INTERVENTIONS:
Biological: EBV-TCR-T Cell Injection — EBV-TCR-T cell injection consists of Epstein-Barr virus-specific T cell receptor-engineered T lymphocytes manufactured from peripheral blood mononuclear cells. These cells are genetically modified to express EBV antigen-specific T cell receptors, enabling targeted recognition and elimination of EBV-infected cells.
  The EBV-TCR-T cells are administered by intravenous infusion at predefined dose levels according to the study protocol, with up to three infusions given at weekly intervals. This intervention is intended to evaluate the safety, tolerability, and preliminary efficacy of EBV-TCR-T cells in patients with EBV DNAemia following allogeneic hematopoietic stem cell transplantation.

SUMMARY:
Epstein-Barr virus (EBV) DNAemia is a common and potentially serious complication after allogeneic hematopoietic stem cell transplantation (allo-HSCT) and may progress to EBV-associated lymphoproliferative disorders. Current treatment options are limited, and effective immune-based therapies are still needed.

This is an investigator-initiated, exploratory, open-label, single-arm clinical study designed to evaluate the safety, tolerability, and preliminary efficacy of EBV-specific T cell receptor-engineered T cells (EBV-TCR-T cell injection) in patients with EBV DNAemia after allo-HSCT. Eligible participants will receive intravenous infusions of EBV-TCR-T cells at escalating dose levels. Safety outcomes, EBV-DNA clearance, and preliminary efficacy will be assessed, along with pharmacokinetic and pharmacodynamic characteristics of the infused cells.

DETAILED DESCRIPTION:
This study is an investigator-initiated, exploratory, open-label, single-arm, dose-escalation clinical trial designed to evaluate the safety, tolerability, and preliminary efficacy of EBV-specific T cell receptor-engineered T cell injection (EBV-TCR-T) in patients with EBV DNAemia following allogeneic hematopoietic stem cell transplantation.

EBV-TCR-T cells are genetically engineered T lymphocytes expressing EBV antigen-specific T cell receptors, enabling targeted recognition and elimination of EBV-infected cells. In this study, peripheral blood mononuclear cells will be collected from the patient or an appropriate donor and used to manufacture EBV-TCR-T cells, which will be administered by intravenous infusion.

The study will enroll approximately 4 to 18 participants. Three dose levels are planned: 1×10^5 cells/kg, 5×10^5 cells/kg, and 1×10^6 cells/kg per infusion. Participants will receive weekly infusions, with up to three infusions administered at Day 0, Day 7, and Day 14, depending on safety and virologic response. Dose escalation will follow a predefined dose-limiting toxicity (DLT)-based design to determine the maximum tolerated dose and the potential optimal biologic dose.

The primary objectives of the study are to evaluate safety and tolerability, including the incidence and severity of adverse events, immune-related adverse events, serious adverse events, and dose-limiting toxicities. Secondary objectives include assessment of preliminary efficacy, such as EBV-DNA clearance rate, time to EBV-DNA negativity, and changes in EBV viral load. Pharmacokinetic and pharmacodynamic analyses will assess in vivo expansion, persistence of EBV-TCR-T cells, and associated immune biomarkers.

Participants will be followed for safety, efficacy, and immune response for up to 12 months after the first infusion, with long-term safety follow-up conducted according to protocol requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of enrollment.
* History of allogeneic hematopoietic stem cell transplantation.
* Presence of Epstein-Barr virus (EBV) DNAemia confirmed by quantitative polymerase chain reaction (qPCR) in peripheral blood.
* EBV DNAemia persisting or increasing despite standard management, as determined by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate organ function as defined by the study protocol.
* Ability to understand and willingness to sign written informed consent.

Exclusion Criteria:

* Diagnosis of EBV-associated lymphoproliferative disorder requiring immediate cytotoxic chemotherapy.
* Active, uncontrolled infection other than EBV.
* History of severe autoimmune disease requiring systemic immunosuppressive therapy.
* Uncontrolled graft-versus-host disease requiring high-dose systemic corticosteroids or other immunosuppressive treatment.
* Prior treatment with EBV-specific adoptive T cell therapy within a defined washout period.
* Known active malignancy other than EBV-related disease that may interfere with study participation.
* Pregnant or breastfeeding women.
* Any medical, psychological, or social condition that, in the opinion of the investigator, would interfere with safe participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of EBV-TCR-T Cell Injection | From the first infusion up to 28 days after the last EBV-TCR-T cell infusion
  Safety and tolerability will be assessed by the incidence, nature, and severity of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) following EBV-TCR-T cell infusion. Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE). Immune-related adverse events, including cytokine release syndrome and other infusion-related reactions, will be closely monitored throughout the study.

SECONDARY OUTCOMES:
EBV DNA Clearance Rate | Up to 3 months after the first EBV-TCR-T cell infusion
  EBV DNA clearance rate is defined as the proportion of participants who achieve EBV DNA negativity in peripheral blood following EBV-TCR-T cell infusion, as measured by quantitative polymerase chain reaction (qPCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns and the sensitive nature of the participant data, individual participant data (IPD) will not be shared. Access to data will be strictly controlled and provided only if required by regulatory authorities.